CLINICAL TRIAL: NCT05514717
Title: A Phase 1, First-in-Human, Dose Escalation and Expansion, Multicenter Study of XMT-2056 in Participants With Advanced/Recurrent Solid Tumors That Express HER2
Brief Title: A Study of XMT-2056 in Advanced/Recurrent Solid Tumors That Express HER2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mersana Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MER-XMT-2056-1
Record Dates: First submitted 2022-08-08; First posted 2022-08-24 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Breast Cancer; HER2-positive Gastric Cancer; HER2-positive Non-Small Cell Lung Cancer; HER2-positive Colorectal Cancer; HER2-positive Tumors; HER2 Low Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- XMT-2056 (Experimental): XMT-2056 alone (monotherapy)
  Interventions: Drug: XMT-2056

INTERVENTIONS:
Drug: XMT-2056 — XMT-2056 will be administered through a vein in your arm or port catheter (intravenously)

SUMMARY:
A Study of XMT-2056 in advanced/recurrent solid tumors that express HER2.

DETAILED DESCRIPTION:
The first-in-human (FIH) study of XMT-2056 is a Phase 1, open-label study of XMT-2056 in previously treated patients with advanced/recurrent solid tumors expressing HER2. The XMT-2056 monotherapy trial will consist of dose escalation (DES) and expansion (EXP) parts.

DES will be the dose-finding portion of the study to assess the safety and tolerability of XMT-2056 and determine the maximum tolerated dose (MTD) and/or Recommended Phase 2 Dose (RP2D). The RP2D will be determined based on the totality of the clinical data, including safety and preliminary anti-tumor effect, PK, and relevant biomarker data.

ELIGIBILITY:
Inclusion Criteria:

* Participant has recurrent or metastatic solid tumors with HER2 expression and has disease progression after treatment, is intolerant to treatment, or is contraindicated with available anti-cancer therapies known to confer benefit, based on investigator's judgement. Note: Participants must have HER2 positivity per the results of their most recent tumor tissue testing, defined as IHC 3+ or IHC 2+ in combination with in situ hybridization (ISH)+. Participants with ERBB2-activating mutations or ERBB2 gene amplification in the absence of HER2 positivity are considered ineligible.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Participant must have measurable disease as defined by RECIST version 1.1.
* Participant has fresh tumor biopsy tissue available for submission to central laboratory. If obtaining fresh tumor tissue is medically contraindicated, archival tumor tissue can be submitted following written approval of the request by the study Medical Monitor. Samples must be obtained after the participant's most recent HER2-targeting therapy unless determined to be medically contraindicated after discussion with the medical monitor.

Exclusion Criteria:

* • Participant is receiving immunosuppressive doses of systemic medications, (doses >10 mg/day prednisone or equivalent) that cannot be discontinued for at least 2 weeks before the first dose and during study drug treatment administration. Note: physiologic hormone replacement therapy is an exception.
* Participant has received prior treatment targeting STING pathway.
* Diagnosis of additional malignancy that required active treatment (including surgery, systemic therapy, and radiation) within the last 2 years, expect for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the breast or the cervix. Participants with an additional malignancy that has a low risk for recurrence may be eligible after discussion with the study Medical Monitor.
* Participants have untreated CNS metastases (including new and progressive brain metastases), history of leptomeningeal metastasis, or carcinomatous meningitis.

  1. Participants are eligible if CNS metastases are adequately treated and participants are neurologically stable for at least 2 weeks prior to enrollment.
  2. In addition, participants must be either off corticosteroids, or on a stable/decreasing dose of ≤ 10 mg prednisone daily (or equivalent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of dose-limiting toxicities (DLTs) associated with XMT-2056 during the first cycle of treatment (Dose Escalation) | 15 months
  Determine the maximum tolerated dose (MTD) of XMT-2056
Incidence of adverse events (Dose Escalation and Dose Expansion) | 3 years
  Assess the safety and tolerability of XMT-2056 by determining the number of patients with adverse events from date of first dose to 30 days post last dose.
Objective Response Rate (ORR) (Dose Expansion) | 3 years
  The percentage of patients with a best overall response of confirmed complete or partial response as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (Dose Escalation) | 3 years
  The percentage of patients with a best overall response of confirmed complete or partial response as assessed by the investigator per Resist Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Duration of response (DOR) (Dose Escalation and Dose Expansion) | 3 years
  The time from when response criteria are first met until disease progression or death in participants who achieve a confirmed complete or partial response.
Disease control rate (DCR) (Dose Escalation and Dose Expansion) | 3 years
  The percentage of patients who achieve a complete response, partial response or stable disease as the result of study treatment
Time of maximum observed plasma concentration of XMT-2056 (Tmax) (Dose Escalation and Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-2056
Maximum observed plasma concentration of XMT-2056 (Cmax) (Dose Escalation and Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-2056
Area under the concentration-time curve of XMT-2056 (AUC) (Dose Escalation and Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-2056
Systemic clearance of XMT-2056 (Dose Escalation and Dose Expansion) | 3 years
  Assess the pharmacokinetics of XmT-2056 by measuring the rate at which the drug is eliminated from the body
Apparent terminal elimination of half-life of XMT-2056 (Dose Escalation and Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-2056
Volume of Distribution (Dose Escalation and Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-2056
Trough concentration of XMT-2056 (Ctrough) (Dose Escalation and Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-2056 by measuring the lowest concentration of drug before dosing
Serum samples for analysis of XMT-2056 antidrug and neutralizing antibodies (ADA/nAb) (Dose Escalation and Dose Expansion) | 3 years
  Assess the development of antidrug antibodies (ADA) and neutralizing antibodies (nAB) to XMT-2056

CONTACTS AND LOCATIONS:
Overall Officials: Brad Sumrow, MD, Study Director — Mersana Therapeutics
Locations (14):
- United States (14):
  - University of South California, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - AdventHealth Celebration, Celebration, Florida
  - Emory Healthcare, Emory Clinic, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York University Medical Oncology Associates, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No